CLINICAL TRIAL: NCT04236388
Title: Short Term Dietary Ketone Drink Consumption and Cardiometabolic Health in Adults
Brief Title: Short Term Ketone Supplementation and Cardiometabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Kevin Davy, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 25-529
Record Dates: First submitted 2020-01-16; First posted 2020-01-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Risk Factor
Keywords: D-β-hydroxybutyrate; low carbohydrate high fat diet; blood pressure; cognitive function; flow mediated dilation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Ketone (Active Comparator): Participants will consume three daily ketone drinks (one before each meal) for 2 weeks.
  Interventions: Dietary Supplement: Ketone drink
- Placebo (Placebo Comparator): Participants will consume three daily placebo drinks (one before each meal) for 2 weeks. .
  Interventions: Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Ketone drink — Pre- and post-testing will be completed before and after participants receive 42 doses of ketone supplement drink over a 2-week period (3x/day for 14 days).
  Arms: Dietary Ketone
Dietary Supplement: Placebo drink — Pre- and post-testing will be completed before and after participants receive 42 doses of placebo supplement drink over a 2-week period (3x/day for 14 days).
  Arms: Placebo

SUMMARY:
The purpose of this research study is to determine if short-term consumption of a dietary ketone drink, which increases the blood circulation concentrations of beta-hydroxybutyrate, a ketone, affects blood vessel health and cognitive health in adults. Ketones are normally produced by the liver when people fast longer than 16-24 hours or eat a diet low in carbohydrates. Participants will be asked to randomly consume a dietary ketone drink and placebo (flavored water) for a 2-week period each in a crossover fashion with a 2-week washout period while maintaining habitual diet and physical activity patterns.

The investigators hypothesize that consumption of a ketone drink will reduce BP and improve vascular health by reducing aortic pulse wave velocity and increasing brachial artery flow mediated dilation. Furthermore, they hypothesize that ketone consumption will improve cognitive health by increasing attention and processing speed.

DETAILED DESCRIPTION:
Objective: The objective of this study is threefold: 1) To establish feasibility and proof-of-concept for the efficacy of ketone supplementation in reducing blood pressure and improving vascular and cognitive function in older adults; 2) Establish proficiency and feasibility with the proposed cognitive function measurements; and 3) Obtain preliminary data for effect size generation.

Background: Age is the primary risk factor for cardiovascular disease. Middle age is a vulnerable period where cardiovascular risk factors, such as BP, begin to emerge and signs and symptoms of disease first becomes evident. Hypertension is present in 60-75% of adults in this demographic and associated with vascular dysfunction and cognitive decline. Low Carbohydrate High Fat (LCHF) ketogenic diets have become increasingly popular for improving cardiometabolic health but adherence is suboptimal due to their restrictive nature. Supplementation with ketone drinks increase plasma β-hydroxybutyrate and mimics the metabolic effects of LCHF ketogenic diets as well as lowers BP and improves vascular and cognitive function in rodent models. Whether ketone supplementation lowers BP and improves vascular and cognitive health in humans of any age is unknown.

Approach: A double-blind randomized 2x2 crossover design with 2 repeated measures in each period will be used. Pre-/post-test evaluation in each period will be used to evaluate the benefits to vascular and cognitive health ingestion with consumption of a ketone drink/placebo drink.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* 50-75 years of age
* Systolic blood pressure <160 mmHg
* Diastolic blood pressure <100 mmHg
* Sedentary to recreationally active
* Body Mass Index <35 kg/m^2
* Postmenopausal women must be >1 year since last menses

Exclusion Criteria:

* Current smoker
* Pregnant or planning to become pregnant
* Dyslipidemia (Total cholesterol >240 mg/dL, LDL >160 mg/dL)
* Chronic clinical disease (e.g., inflammatory bowel disease/irritable bowel syndrome, unstable coronary heart disease, stroke, heart failure, diabetes, neurological disorders)
* Following an extreme dietary pattern or planning to change to one (e.g., low carbohydrate, carnivore)
* Not weight stable in the prior 3 months (>2 kg weight change)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Change in Arterial Stiffness after Supplementation | 45-minute measurement in laboratory
  The blood flow and diameter in the common arteries in the neck will be measured from the image obtained from an ultrasound unit (GE Vivid S6) equipped with a high-resolution linear array transducer. For applanation tonometry, the carotid, brachial, radial and femoral artery pressure waveform and amplitude will be obtained by a fingertip probe incorporating a high-fidelity strain gauge transducer. Each of these measures are used to calculate arterial stiffness. These tests will be conducted two times separated by about 2 weeks. The participant will be randomly-assigned to a supplement drink (ketone or placebo) followed by a 2-week washout period (crossover design). The supplement drink will be consumed 3 times per day, once before each meal.
Change in Brachial Artery Function after Supplementation | 30-minute measurement in laboratory
  Brachial artery function or flow mediated dilation (FMD), the blood flow and diameter of the brachial artery in the forearm (fMD), will be measured using a duplex ultrasound machine before and after the inflation of a blood pressure cuff on the forearm for 5 minutes and after placing a nitroglycerine tablet (0.4 mg) under the participant's tongue. This test will be conducted two times separated by about 2 weeks. The participant will be randomly-assigned to a supplement drink (ketone or placebo) followed by a 2-week washout period (crossover design). The supplement drink will be consumed 3 times per day, once before each meal. Off-line analysis of baseline and post-reactive hyperemic diameters and velocities will be performed using edge detection software (Vascular Analysis Tools, Medical Imaging Applications, Inc.).

SECONDARY OUTCOMES:
Change in Blood Pressure after Supplementation | 15-minute measurement in laboratory
  Blood pressure measurements will be made under quiet, comfortable ambient laboratory conditions via mercury sphygmomanometry. Three consecutive measurements within 6mmHg will be averaged. This measurement will be conducted two times separated by about 2 weeks. The participant will be randomly-assigned to a supplement drink (ketone or placebo) followed by a 2-week washout period (crossover design). The supplement drink will be consumed 3 times per day, once before each meal.
Change in Glucose Tolerance after Supplementation | 2-hour test in laboratory
  Participants will complete an oral glucose tolerance test, which includes having each subject consume a sugary glucose drink (75 grams) and collecting small amounts (less than one half teaspoon) of blood every half hour (4 blood draws) for a 2-hour period. These tests will be conducted two times separated by about 2 weeks. Each participant will be randomly-assigned to a supplement drink (ketone or placebo) followed by a 2-week washout period (crossover design). The supplement drink will be consumed 3 times per day, once before each meal.
Change in 24-hour Area Under the Curve for Glucose Levels after Supplementation | 3-day measurement during free living
  Glucose will be monitored by a Continuous Glucose Monitor (CGM) sensor (Enlite Sensor, Medtronic, Inc. or FreeStyle Libre, Abbott) and this will be placed on the subject's abdomen or back of the upper arm in order to measure glucose continuously. The measured glucose levels will be assessed by an iPro2 Professional CGM, Medtronic, Inc. or FreeStyle Libre Pro CGM, Abbott and the CGM will be worn for consecutive 3 days. These tests will be conducted two times separated by about 2 weeks. The participant will be randomly-assigned to a supplement drink (ketone or placebo) followed by a 2-week washout period (crossover design). The supplement drink will be consumed 3 times per day, once before each meal.
Change in Executive Cognitive Function after Supplementation | 40-min measurement in laboratory
  Participants will be instructed to complete a set of computerized tasks to asses executive cognitive function (e.g., working memory), speed of processing, and semantic verbal fluency. These tests will be conducted two times separated by about 2 weeks. The participant will be randomly-assigned to a supplement drink (ketone or placebo) followed by a 2-week washout period (crossover design). The supplement drink will be consumed 3 times per day, once before each meal.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Davy, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Polytechnic and State University, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No